CLINICAL TRIAL: NCT03724071
Title: A Phase I/IIa Study of TG6002 (VV TK-RR-FCU1) Administered by Intravenous (IV) Infusions in Combination With Oral Flucytosine (5-FC) in Patients With Advanced Gastro-intestinal (GI) Tumors.
Brief Title: Study of TG6002 (VV TK-RR-FCU1) in Combination With 5-FC in Patients With Advanced Gastro-intestinal Tumors.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study has been terminated after Phase I part on 23 February 2023
Sponsor: Transgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG6002.02
Record Dates: First submitted 2018-10-16; First posted 2018-10-30 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Neoplasm; Digestive System Neoplasm
MeSH Terms: conditions — Colorectal Neoplasms; Digestive System Neoplasms | interventions — Flucytosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1, Arm A - Dose escalation and safety of TG6002 and flucytosine combination (Experimental): Dose escalation with repeated administrations of TG6002 in combination with flucytosine in patients with advanced gastro-intestinal (GI) tumors.
  Interventions: Biological: TG6002; Drug: Flucytosine (5-FC, Ancotil)
- Phase 1, Arm B - Dose escalation and safety of TG6002 and flucytosine combination (Experimental): Dose escalation with closer administrations of TG6002 in combination with flucytosine in patients with advanced gastro-intestinal (GI) tumors.
  Interventions: Biological: TG6002; Drug: Flucytosine (5-FC, Ancotil)
- Phase IIa - Efficacy of TG6002 and flucytosine combination (Experimental): Repeated administrations of TG6002 in combination with flucytosine in patients with colorectal cancer and liver metastases
  Interventions: Biological: TG6002; Drug: Flucytosine (5-FC, Ancotil)

INTERVENTIONS:
Biological: TG6002 — Phase I, Arm A: Dose escalation from 1 x 10E6 PFU to 1 x 10E9 PFU; Phase I, Arm B: Dose escalation from 1 x 10E9 PFU to 1 x 10E10 PFU; Phase II: Established recommended Phase II dose (RP2D)
  Administration intravenously on Days 1, 8 and 15 (Phase I, Arm A) or on Days 1, 3 and 5 (Phase I, Arm B). Three intravenous infusions at the Dose Recommended for Phase 2 (RP2D) in Phase IIa.
  An extension of the 28-day cycle of TG6002/5-FC combination can be repeated in case of evidence of patient benefit, defined as an objective radiological response or disease stabilization, and/or a clinically significant relief in patient's symptoms. Additional cycle(s) will start from 2 to 4 weeks following the last 5-FC intake.
Drug: Flucytosine (5-FC, Ancotil) — Administered orally at a dose of 200 mg/kg/day for a total of 10 days (Phase I, Arm B) or 16 days (Phase I, Arm A).
  An extension of the cycle of TG6002/5-FC combination can be repeated in case of evidence of patient benefit, defined as an objective radiological response or disease stabilization, and/or a clinically significant relief in patient's symptoms.

SUMMARY:
This study will include two parts:

* In the phase I part: safety will be assessed in consecutive cohorts of 3 to 6 patients at increasing doses of TG6002 in combination with oral flucytosine (5-FC) in patients with advanced gastro-intestinal (GI) tumors.
* In the phase IIa part: evaluation of efficacy and further evaluation of safety of multiple administrations of TG6002 in combination with flucytosine (5-FC) in patients with colorectal cancer and liver metastases.

In both parts, tumor response will be evaluated on local assessment using RECIST 1.1.

All patients will be followed up until disease progression or death due to any cause or the date of data cut-off, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Patient population:

   * Phase I part: patients with advanced GI carcinomas having failed and/or intolerant to standard therapeutic options. Patients must have been previously exposed to fluoropyrimidine-based chemotherapy.
   * Phase IIa part: patients with colorectal cancer and liver metastases having failed and/or intolerant to standard therapeutic options. Standard treatment consists of fluoropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy, possibly combined with an anti-VEGF and/or an anti-EGFR monoclonal antibody. In addition, the patient should not be candidate to a treatment with regorafenib.
2. Male or female aged ≥18 years.
3. a. Patient presenting with at least one measurable lesion according to RECIST 1.1 in Phase IIa part (optional in the Phase I part) b. Patient presenting with at least one biopsiable metastatic non target lesion (liver metastasis in the Phase IIa part)
4. Expected survival of at least 12 weeks
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
6. Absolute neutrophil count (ANC) ≥1000/mm3
7. Blood lymphocyte count ≥500/mm3
8. Hemoglobin (Hb) level ≥10 g/dL
9. Platelet count ≥100,000/mm3
10. Total bilirubin ≤1.5 x Upper Limit of Normal (ULN), except patients with Gilbert syndrome who must have a total bilirubin level of <3.0 x ULN
11. AST, ALT, alkaline phosphatase ≤3 x ULN, unless if liver metastases are present (≤5 x ULN in that case)
12. Clearance for study participation and anti-hypertensive therapy suspension (see exclusion criterion 13) after cardiology consultation and cardiologic investigations including troponin T or I blood level, electrocardiogram (ECG) and cardiac echography (ECHO)
13. Negative blood pregnancy test for women of childbearing potential (WOCBP)
14. Highly effective method of contraception (i.e. methods with a failure rate of less than 1% per year) combined with a barrier method (e.g. condom) for male and female patients during TG6002 treatment period and for a minimum of 3 months following the last administration of TG6002
15. Signed written informed consent in accordance to ICH-GCP and national/local regulation

Exclusion Criteria:

1. Previous irradiation of target tumor
2. MSI-High/dMMR colorectal cancer patients
3. Glomerular filtration rate <60 mL/min/1.73m2 according to the Modification of Diet in Renal Diseases (MDRD) formula
4. Immunodeficiency due to underlying illness (e.g. HIV/AIDS) and/or immunosuppressant agent, including systemic corticosteroids at a dose >10 mg/day of equivalent prednisolone taken for more than 4 weeks within 3 months prior to TG6002 treatment initiation
5. History of severe exfoliative skin condition (e.g. eczema or atopic dermatitis) requiring systemic therapy for more than 4 weeks within 2 years prior to TG6002 treatment initiation
6. Significant impairment of GI tract absorption, such as total gastrectomy, gastric mucosal atrophy, extensive intestinal resections or malabsorption disease
7. Symptomatic bacterial intestinal overgrowth consecutive to intestinal dysmotility, surgical resections (blind loops, ileo-cecal valve), or anatomical abnormalities
8. Inflammatory bowel disease (IBD) requiring treatment within the past 2 years prior to TG6002 administration and bowel sub-obstruction
9. Known deficiency in dihydropyrimidine dehydrogenase (DPD)
10. Known hypersensitivity to 5-FC or its excipients
11. Known hypersensitivity to eggs or gentamycin
12. Severe or unstable cardiac disease, including significant coronary artery disease (e.g. requiring angioplasty or stenting) within 12 months prior to TG6002 treatment initiation, unless well-controlled and on stable medical therapy for at least 6 months
13. Inability to withdraw anti-hypertensive therapy 24 hours prior to and up to 24 hours after TG6002 treatment AND/OR patients treated with 3 or more anti-hypertensive agents AND/OR patients with signs of advanced hypertensive disease, such as renal function impairment, left ventricular hypertrophy, hypertensive encephalitis or history of hemorrhagic stroke
14. Patients with other malignancies than the target disease in this trial except cutaneous basal cell carcinoma and in situ carcinoma of the uterine cervix, unless complete remission for at least 5 years prior to study entry and no additional therapy required during the study
15. Systemic anti-cancer therapy or resection surgery within 4 weeks prior to first administration of TG6002
16. Prior participation in another clinical study involving an IMP with last intake within 4 weeks prior to TG6002 treatment initiation
17. Other medical condition or laboratory abnormality that in the judgment of the investigator may increase the risk associated with study participation or may interfere with interpretation of study results
18. Prior gene therapy
19. Concurrent antiviral therapy active on vaccinia viruses (e.g. ribavirin)
20. Nursing (e.g. lactating) females
21. History of severe systemic reaction or side-effect after a smallpox vaccination, such as systemic vaccinia, eczema vaccinatum, encephalitis, myocarditis, pericarditis
22. Any psychological, familiar, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
23. Patient unable or unwilling to comply with the protocol requirements
24. Severe uncontrolled coagulopathy OR anticoagulant medication for therapeutic purposes that cannot be discontinued prior to liver metastasis or other deep-seated tumor biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Phase I part - Dose-limiting toxicities | Day 28
  Dose-limiting toxicities
Phase II part - Overall response rate | Day 43
  Overall response rate according to Recist v1.1

CONTACTS AND LOCATIONS:
Locations (7):
- Institut Jules Bordet, Brussels, Belgium
- France (2):
  - Centre Léon Bérard, Lyon
  - IUCT Toulouse, Toulouse
- Spain (4):
  - Centro Integral Oncológico Clara Campal (CIOCC) Hospital, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Instituto de Investigación Sanitaria Fundación Jimenez Díaz, Madrid
  - Hospital Clinico Universitario, Valencia

IPD SHARING:
Plan to Share IPD: Undecided